CLINICAL TRIAL: NCT02947282
Title: PREgnancy-associated Pelvic Floor Health Knowledge And REDuction of Symptoms: The PREPARED Trial
Acronym: PREPARED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H12-03450
Record Dates: First submitted 2016-10-11; First posted 2016-10-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Pelvic Organ Prolapse, Patient Education
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Educational Workshop
  Interventions: Other: Educational Workshop
- Control (No Intervention): They will continue regular prenatal care as planned

INTERVENTIONS:
Other: Educational Workshop — They will attend a 2 hour class on pelvic floor health
  Arms: Intervention

SUMMARY:
The pelvic floor is composed of muscles and connective tissue which acts to provide support for pelvic organs, and weakness or injury to the pelvic floor can result in pelvic floor dysfunction. Respect for patient autonomy is a guiding principle in medicine and is of increasing importance for patients. The PREPARED Trial hopes to demonstrate whether a single workshop on pelvic floor health during pregnancy will lead to improved knowledge of pelvic floor symptoms postpartum, increase the practice of pelvic floor muscle exercises, increase satisfaction with their delivery experience, and change participants preferences and thoughts surrounding various modes of delivery.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to determine if a single class on pelvic floor health administered during pregnancy will increase primiparous women's knowledge of pelvic floor health, decrease pelvic floor symptoms postpartum, increase the practice of pelvic floor muscle exercises, increase satisfaction with their delivery experience, and change their preferences and thoughts surrounding various modes of delivery. There are currently no such workshops being provided at St. Paul's Hospital in Vancouver BC.

Hypothesis or Aim: A single 2 hour workshop on pelvic floor health administered during pregnancy will improve primiparous women's knowledge of pelvic floor health at 6 weeks postpartum compared to a control group who do not participate in the workshop.

Justification of the Study (Background): The pelvic floor is composed of muscles and connective tissue which act to provide support for pelvic organs. Weakness or injury to the pelvic floor can result in pelvic floor dysfunction. This includes conditions such as pelvic organ prolapse, urinary incontinence, irritative bladder symptoms, fecal incontinence, pelvic pain and sexual dysfunction. Maintenance of pelvic floor health is important as diseases of the pelvic floor are bothersome, disfiguring and significantly affect quality of life of women. Though the prevalence of pelvic floor problems increases with age, it also affects women of childbearing age, especially during and after pregnancy. According to Brown et al., the prevalence of urinary incontinence 12 months before pregnancy was 10.8% and this increased to 55.9% in the third trimester. At three months postpartum, 30% of women continue to have urinary incontinence. Parity has been strongly associated with pelvic floor dysfunction later in life. According to Rortveit et al, the risk of pelvic organ prolapse was significantly increased in women with 1 (OR 2.8, 95% CI 1.1-7.2), 2 (OR 4.1, 95% CI 1.8-9.5) and 3 or more (OR 5.3, 95% CI 2.3-12.3) vaginal deliveries compared with nulliparous women. Also, forceps delivery has been associated with an increase in pelvic floor symptoms 5-10 years after delivery, especially overactive bladder (OR 2.92, 95% CI 1.44-5.93) and prolapse (OR 1.95, 95% CI 1.03-3.70).

Research on pelvic floor health education by the principal investigator showed that with improvement of pelvic floor health knowledge, there was also improvement in pelvic floor symptoms and quality of life at 3 months after a single workshop. However, introduction of pelvic floor health through a workshop would be ideal in the pregnant population, as they are a captive audience. This is the time when they employ other interventions to improve their health, such as smoking cessation, vitamin supplementation, healthy eating etc. Also, women of childbearing age are of the millennial generation. They have more interest in their own health and place greater value on quality of life compared to previous generations. Thus they are a group of motivated individuals who would implement changes to improve their future quality of life if given the appropriate information to encourage this change.

Despite current evidence demonstrating that the single most important risk factor for disruption of pelvic floor health is childbirth, pregnant women are ill-informed about pelvic floor health. A survey of health professionals in Swansea, UK, revealed that pelvic floor muscle exercises and pelvic floor health received low priority in comparison to other antenatal topics discussed by obstetric care providers with their patients. What is perhaps even more astounding was the finding that 15% of respondents, which included obstetricians, midwives and family physicians, were unable to describe pelvic floor exercises, and most health professionals surveyed felt that they had not received adequate training on pelvic floor health.

Canada does not currently have recommendations on patient education regarding pelvic floor health during pregnancy. As demonstrated by the audit performed by Ismail et al., even in a region where these guidelines exist, the education of pregnant women on this subject is poor. Our current standard of practice is to leave pelvic floor education in the hands of obstetric care providers. A survey of health professionals in the UK revealed that pelvic floor health received low priority in comparison to other topics discussed in the antenatal period. Furthermore, most obstetric care providers felt their training in pelvic floor health was inadequate. The investigators research project proposes to close the gap between patient knowledge and scientific knowledge. There is clear evidence that childbirth is the single most important risk factor in future pelvic floor conditions. There is also evidence in support of pelvic floor muscle exercises in the antepartum and postpartum period to prevent and improve pelvic floor symptoms. The investigators workshop will empower women with knowledge and allow them to make informed decisions surrounding childbirth. It will provide them with tools to improve their own pelvic floor health. A pelvic floor health workshop in the antenatal period is an innovative concept which could lead to better patient care. It may be the first step in prevention of future pelvic floor conditions.

The target population is primiparous women, 20 years or older in their first pregnancy and singleton gestation with 100 women being recruited.

Sampling method: All participants will be randomized to two groups, the random allocation lists will be generated by a statistician unassociated with the study using the SAS programming language. The allocations will be loaded onto a computer and access by a study coordinator interacting with a web-based ORACLE screen. Interactions between the coordinator and the system will be logged, including the time and date, a patient identifier (patient letter code) and the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Women 20 years or older, in their first pregnancy, singleton gestation, from various obstetrical care providers (general practitioner, midwife, obstetrician), planning to deliver at St. Paul's hospital in Vancouver

Exclusion Criteria:

* Women under 20 years of age, multiple gestation, unable to understand English

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Difference in scores on a pelvic floor knowledge questionnaire at 6 weeks postpartum between intervention and control groups | At 6 weeks post-partum

SECONDARY OUTCOMES:
Difference in Pelvic Floor Distress Inventory questionnaire scores at 6 weeks postpartum between intervention and control groups | At 6 weeks postpartum
Difference in questionnaire scores based on Pelvic Floor Knowledge questionnaire postpartum between intervention and control groups | At 6 weeks postpartum
Difference in questionnaire scores on Pelvic Floor Impact Questionnaire between intervention and control groups at 6 weeks postpartum. | At 6 weeks postpartum
Difference in knowledge of practice of pelvic floor muscle exercises based on postpartum questionnaire scores at 6 weeks postpartum between intervention and control groups based on postpartum questionnaire | At 6 weeks postpartum
Difference in frequency of practice of pelvic floor muscle exercises based on postpartum questionnaire scores at 6 weeks postpartum between intervention and control groups based on postpartum questionnaire | At 6 weeks postpartum
Change in mode of delivery preferences before and after the class in the intervention group based on the postpartum questionnaire. | At Delivery
Difference in actual mode of delivery between intervention and control groups based on the postpartum questionnaire | At Delivery
Difference in global satisfaction rating with pelvic floor health and mode of delivery at 6 weeks postpartum between intervention and control groups based on postpartum questionnaire | At 6 weeks post partum

CONTACTS AND LOCATIONS:
Locations (1):
- Nicole Koenig, Vancouver, British Columbia, Canada